CLINICAL TRIAL: NCT02635256
Title: Hypofractionated Radiosurgery for Localised Prostate Cancer
Acronym: HYPOSTAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Luebeck (Other); Saphir Radiosurgery Center Northern Germany (Unknown)
Responsible Party: Principal Investigator, Juergen Dunst, Prof., Prof. Dr. med. Juergen Dunst, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZKS-121-003; ARO-2016-5 (Other: German Cancer Society)
Record Dates: First submitted 2015-12-08; First posted 2015-12-18 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: hypofractionation; prostate cancer; radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypofractionated Radiosurgery (Experimental): 5 fractions with 7 Gy, total dose 35 Gy
  Interventions: Radiation: Hypofractionated Radiosurgery

INTERVENTIONS:
Radiation: Hypofractionated Radiosurgery — Image-guided stereotactic Linac based RT preferable with "dedicated radiosurgery system" such as CyberKnife

SUMMARY:
Hypofractionated radiosurgery has been investigated in a few trials and appears to be safe and feasible.

Investigators initiated this multicenter phase II prospective trial to analyse feasibility (toxicity) of hypofractionated radiosurgery with 5 fractions in patients with localised prostate cancer, who are ineligible for the "PREFERE trial" under the hypothesis that the ratio of patients with late toxicity ≥ grade 2 after 1 year amounts 2,8% and is significant lower than 17.5%.

DETAILED DESCRIPTION:
Experimental radiosurgery of prostate with 5 fractions each with 7,00 Gy (total application rate of 35,00 Gy).

Planned visits are: Baseline, visits at every radiation day and four follow ups (4-6 weeks, 3 months, 6 months and one year after last day of radiation).

ELIGIBILITY:
Inclusion Criteria:

* Localised, histopathologically confirmed Prostate Cancer (cT1-3 N0 M0)
* Gleason-grade ≤7
* Guideline-based staging
* Age ≥ 60 years
* PSA < 15 ng/ml
* Volume of the prostate <80 cm³
* IPSS-Score ≤12
* Written informed consent

Exclusion Criteria:

* History of prior pelvic radiotherapy
* Contraindication to MRI or Fiducial marker implantation (e.g. allergy to gold),
* Immunosuppressive therapy
* Relevant comorbidity thought to adversely affect treatment compliance,
* Legal incapacity or lack of informed consent

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Late toxicity measured with Radiation Therapy Oncology Group-(RTOG)-Score | 12-15 months after radiotherapy

SECONDARY OUTCOMES:
Acute toxicity analysed by Adverse Event (AE)- and Serious Adverse Event (SAE)-reports. | through study completion
Prostate Specific Antigen (PSA) | At the time of inclusion and 1, 3, 6-9 and 12-15 months after radiotherapy
International Prostate Symptom Score (IPSS) | Screening and 3, 6-9 and 12-15 months after radiotherapy
EORTC Quality of Life Questionnaire (QLQ) C30 | At the time of inclusion and 12-15 months after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Dunst, Prof., Principal Investigator — University Hospital Schleswig-Holstein
Locations (5):
- Germany (5):
  - Saphir Radiosurgery Center Frankfurt am Main, Frankfurt am Main
  - University Hospital Frankfurt, Department of Radiation Therapy and Oncology, Frankfurt am Main
  - Saphir Radiosurgery Center Northern Germany, Güstrow
  - University Medical Center Schleswig-Holstein, Kiel
  - European Cyberknife Center Munich, Munich

REFERENCES:
- [Background] Jiang P, Krockenberger K, Vonthein R, Tereszczuk J, Schreiber A, Liebau S, Huttenlocher S, Imhoff D, Balermpas P, Keller C, Dellas K, Baumann R, Rodel C, Hildebrandt G, Junemann KP, Merseburger AS, Katz A, Ziegler A, Blanck O, Dunst J. Hypo-fractionated SBRT for localized prostate cancer: a German bi-center single treatment group feasibility trial. Radiat Oncol. 2017 Aug 18;12(1):138. doi: 10.1186/s13014-017-0872-2. PMID 28821268
- [Result] Krug D, Imhoff D, Haidenberger A, Hessler N, Schafer J, Huttenlocher S, Chatzikonstantinou G, Furweger C, Ramm U, Konig IR, Chun F, Staehler M, Rodel C, Muacevic A, Vonthein R, Dunst J, Blanck O. Robotic stereotactic body radiotherapy for localized prostate cancer: final analysis of the German HYPOSTAT trial. Strahlenther Onkol. 2023 Jun;199(6):565-573. doi: 10.1007/s00066-023-02044-2. Epub 2023 Feb 9. PMID 36757424